CLINICAL TRIAL: NCT01140087
Title: Maxillofacial Composite Tissue Allograft Transplantation: Face Transplant
Brief Title: Face Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Rolf Barth, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040219; N00014-07-1-0298 (Other Grant/Funding Number: ONR)
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Transplantation: Facial Transplantation
Keywords: Face Transplant; Composite Tissue Allograft; Facial Allotransplantation
MeSH Terms: interventions — Facial Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional (Experimental): Face Transplantation
  Interventions: Procedure: Face Transplant

INTERVENTIONS:
Procedure: Face Transplant — Transplantation of donor facial skin, tissue, muscle, and bone as needed

SUMMARY:
This study aims to:

1. Perform face transplants on people who have suffered severe facial trauma with tissue and functional loss; and
2. Evaluate the acceptance and function of the transplanted tissue.

DETAILED DESCRIPTION:
For patients with severe facial deformities or facial wounds from traumatic injuries, we would like to pursue the use of a face transplant to help reconstruct a person's damaged face. Our goal is to not only give the patient back a normal appearance to their face but also the functioning, movement, and sensation of their face including that of the lips, mouth, and eyes. For some patients with severe face deformities simple tasks such as smiling, talking, eating, kissing a loved one, or even just being able to contain their saliva become difficult, if not impossible. These patients often become depressed because of their facial deformities.

Although there are some techniques in plastic and reconstructive surgery that can repair the look of a patient's face, often these cannot replace the moving parts of the face. Currently, patients with severe facial deformities would undergo several reconstructive surgeries with their own tissues, called autologous transplant. This surgery often leaves unacceptable scars and deformities of the patient's donor sites. Also, this conventional reconstruction method requires many returns to the operating room to carefully form and shape the transplanted free flap. Lastly, this type of reconstruction is still limited, as it does not provide a reliable return in function, sensation, and appearance for the damaged parts of the face.

Instead, if we use a composite tissue allograft (CTA), or face transplant from a donor who is brain dead such as in heart, kidney and liver transplants, we could replace the damaged parts of the face with the same missing parts that could return movement as well. However, since the transplanted facial tissues are from another person, these face transplant recipients need medicines that would keep their body from rejecting the new tissues. This new course of medicines would be their daily responsibility. Though there are risks with taking these medicines, the risks have been lowered by many prior studies that have been done with patients who have had other organ transplants. However, the risks are still a consideration when deciding to choose this option for correcting severe facial deformities.

This study aims to perform a face transplant on a person who has suffered a severe facial trauma with tissue and functional loss, and with limited other established surgical options to repair their deformities. We will conduct the surgery and prospectively follow the patient to monitor his or her clinical and functional outcomes and ensure that optimal results are achieved. We will systematically document and record the entire process of the patient's surgery and recovery. An important factor of this surgery's success is that the patient strictly follows and takes the required course of medicines to prevent rejection of the donor tissues. In order to ensure that the tissue survives and is not rejected by the patient, we will continuously check various clinical values, such as blood work, tissue samples, and x-ray images.

We would like to offer facial segment transplantation as a reconstructive option to patients with severe facial deformities. We feel facial transplantation has now become a viable option for certain patients. If successful, this will contribute to future research and development in the field of tissue transplantation. Most importantly, our goal is to offer patients the best option in reconstruction to restore both form and function who otherwise do not have another option.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* Facial defect or injury requiring facial transplantation as determined by the treating Plastic and Reconstructive Surgeon
* Signed written informed consent
* Able to complete psychiatric evaluations
* Willing and able to continue immunosuppression regimen as directed by treating physician
* Willing and able to return for follow-up visits as described in the treatment plan
* Must have autogenous tissue options available for reconstruction in event of graft failure
* Laboratory values as defined by research protocol
* Willing to undergo review by Participant Selection Committee and be placed on a transplant recipient waitlist

Exclusion Criteria:

* Pre-existing disease that would exclude the recipient from transplantation
* Active infection
* Ongoing substance abuse
* HIV positive
* Positive for Hepatitis B or C
* Active malignancy
* Pregnant or breastfeeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-09; Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Evaluate the success of the face transplant | Monthly for 6 months, every 6 months for 2 years, then annually
  We will measure the restoration of function, sensation, and appearance of the transplanted facial segment

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Barth, MD, Principal Investigator — U of Maryland
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States